CLINICAL TRIAL: NCT01222039
Title: Multicenter Clinical Trial Phase I/II Randomized, Controlled, for the Evaluation of Safety and Feasibility of Therapy With Two Different Doses of Allogenic Mesenchymal Stem Cells From Adipose Tissue in Patients With Chronic Graft Versus Host Disease.
Brief Title: Multicenter Clinical Trial for the Evaluation of Mesenchymal Stem Cells From Adipose Tissue in Patients With Chronic Graft Versus Host Disease.
Acronym: CMM/EICH/2008
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2008-004014-27
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Graft Versus Host Disease; Chronic and Expanded Graft Versus Host Disease; Immune System Diseases
Keywords: Graft versus host disease; Mesenchymal stem cell; Allogeneic mesenchymal stem cell; Adipose tissue; Allotransplant; Allogenic; Mesenchymal Stem Cells; Immune System Diseases; Chronic; Expanded
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional treatment plus high dose: 3x10e6 cells / Kg. (Experimental): Conventional treatment:Gradually descending dosage of prednisone and cyclosporin or tacrolimus for at least 46 weeks. Starting dose: 1 mg/Kg/24 h prednisone and 3 mg/Kg/12 h cyclosporin.
  Interventions: Other: Conventional treatment plus intravenous infusion of allogenic mesenchymal stem cells from adipose tissue.
- Conventional treatment plus low dose: 1x10e6 cells / Kg (Experimental): Conventional treatment:Gradually descending dosage of prednisone and cyclosporin or tacrolimus for at least 46 weeks. Starting dose: 1 mg/Kg/24 h prednisone and 3 mg/Kg/12 h cyclosporin.
  Interventions: Other: Conventional treatment plus intravenous infusion of allogenic mesenchymal stem cells from adipose tissue.

INTERVENTIONS:
Other: Conventional treatment plus intravenous infusion of allogenic mesenchymal stem cells from adipose tissue. — Conventional treatment plus intravenous infusion of allogenic mesenchymal stem cells from adipose tissue. Low dose: 1 x10e6 / Kg.
  Conventional treatment:Gradually descending dosage of prednisone and cyclosporin or tacrolimus for at least 46 weeks. Starting dose: 1 mg/Kg/24 h prednisone and 3 mg/Kg/12 h cyclosporin.
Other: Conventional treatment plus intravenous infusion of allogenic mesenchymal stem cells from adipose tissue. — Conventional treatment plus intravenous infusion of allogenic mesenchymal stem cells from adipose tissue. High dose: 3 x10e6/Kg.
  Conventional treatment:Gradually descending dosage of prednisone and cyclosporin or tacrolimus for at least 46 weeks. Starting dose: 1 mg/Kg/24 h prednisone and 3 mg/Kg/12 h cyclosporin.

SUMMARY:
The main purpose of this trial is to assess the safety and feasibility of treatment with two-dose infusion of allogeneic mesenchymal stem cells from adipose tissue expanded in vitro in patients undergoing haematopoietic stem cell transplantation (HSCT, who have developed chronic and extensive graft versus host disease (GVHD).

Mesenchymal stem cells (MSCs) express low levels of HLA class I molecules, and do not express class II molecules neither CD40, CD80 and CD86, being unable to induce proliferation of allogeneic lymphocytes. In addition, MSCs inhibit lymphocyte proliferation by inhibiting cell division and maintaining these cells in a quiescent state. This supports the hypothesis that MSCs are universal suppressors.

ELIGIBILITY:
Inclusion Criteria:

Patients who develop chronic extensive GVHD as determined by the National Institute of Health Consensus Development Project on Criteria for Clinical Trials in Chronic GVHD (Biol Blood Marrow Transplant 2005; 11: 945-955), and which meet the following criteria:

1. They have never received therapy for chronic GVHD.
2. They have de novo or quiescent chronic extended GVHD.

Exclusion Criteria:

1. Concomitant severe systemic infection.
2. Oncologic or hematological condition relapse.
3. Pregnancy.
4. Estimated life expectancy less than 1 week.
5. Patients who do not give their informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 24 months

SECONDARY OUTCOMES:
Percentage of patients in each group that may potentially reduce corticosteroids at week 7, 20 and 42, started immunosuppressive treatment and percentage of patients at week 56 have been suspended on full immunosuppressive treatment | 12 months
Overall survival and disease-free survival. | 12 months
Changes in lymphocyte subsets and levels of inflammatory and antiinflammatory cytokines in each of the groups. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Jurado Chacón, MD, Study Chair — Haematology Department, Hospital Universitario Virgen de las Nieves de Granada. Spain.; Ildefonso Espigado, MD, Principal Investigator — Haematology Department, Hospital Universitario Virgen del Rocío de Sevilla, Spain.; Carlos Solano Vercet, MD, Principal Investigator — Haematology and Oncology Department. Hospital Clínico Universitario de Valencia, Spain.; Sebastián Garzón López., MD, Principal Investigator — Hospital de Jerez de la Frontera, Cádiz. Spain.
Locations (4):
- Spain (4):
  - Hospital de Jerez de la Frontera., Jerez de la Frontera, Cádiz.
  - Hospital Universitario Virgen de las Nieves, Granada, Granada.
  - Hospital Universitario Virgen del Rocío de Sevilla, Seville, Sevilla
  - Hospital Clínico de Valencia, Valencia, Valencia